CLINICAL TRIAL: NCT04174898
Title: Human Mesenchymal Stem Cell (hMSC) Infusion for Anti-Aging and REGENerative Therapy
Brief Title: MSC Infusion for Anti-aging and Regenerative Therapy
Acronym: REGEN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Landmark Medical Centre Sdn Bhd (Other)
Collaborators: CytoMed Therapeutics Pte Ltd (Industry)
Responsible Party: Principal Investigator, Dr Lucas Luk Tien Wee, Director, Consultant Obstetrician & Gynaecologist, Landmark Medical Centre Sdn Bhd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Protocol LMC-101
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Aging Well; Regenerative Medicine
Keywords: human Mesenchymal Stem Cells (hMSC); Anti-Aging; Regenerative Medicine; Adipose Derived MSCs; Umbilical Cord Derived MSCs; Autologous hMSC; Allogenic hMSC

STUDY DESIGN:
Intervention Model Description: Prospective, Unblinded, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Population (Experimental): 100 million human MSCs in 200mls of normal saline, intravenously, once-off, over 1-2hours
  Interventions: Biological: human Mesenchymal Stem Cell (MSC) infusion therapy

INTERVENTIONS:
Biological: human Mesenchymal Stem Cell (MSC) infusion therapy — Subjects will be infused with 100million human MSCs

SUMMARY:
To evaluate the safety and efficacy of human Mesenchymal Stem Cell (hMSC) infusion therapy, in preserving general wellness and ameliorating or reversing the effects of aging in our study population

DETAILED DESCRIPTION:
100million human mesenchymal stem cells will be infused into study subjects. They will be followed up for both objective and subjective measures of 'anti-aging'. Biochemical markers such as male and female hormones and other parameters of well being will be measured. A questionnaire will also be filled pre and post infusion to ascertain one's well-being (Adapted from SF-36).

Source of MSCs - Autologous (Adipose tissue) or Allogenic (Adipose tissue or umbilical cord)

MSC production and storage will be performed in a GMP certified laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

1. All patients >18yrs old, who are able to read, write and understand Informed Consent form, regarding the experimental nature of this therapy.
2. All Healthy Subjects are eligible for this study
3. Subjects with stable pre-morbid medical conditions, not requiring changes to their current medical therapy for >6 months prior to enrolling in this study, are eligible.

Exclusion Criteria:

1. Uncontrolled blood pressure at the time of enrollment: systolic pressure >160 mmHg and/or diastolic blood pressure > 100 mmHg.
2. Having evidence related to renal dysfunction: creatinine > 1.5 mg/dl or (>133 mmol/L) for men. creatinine > 1.4 mg/dl or (>124 mmol/L) for woman. eGRF < 40 ml/ min Proteinuria > 300 mg/day
3. Severe heart disease (NYHA 3/4 or congestive heart failure)
4. Severe liver disease (liver enzymes >2x baseline, or evidence of coagulopathy)
5. Evidence of ketoacidosis at the time of selection.
6. Evidence of ongoing or frequent hypoglycemia.
7. Severe infection at time of selection
8. Infected with hepatitis B virus or hepatitis C or tuberculosis.
9. Serious allergic constitution
10. Neoplasm detected before/during screening or raised tumour markers CA125 (Females), CA15.3 (Females), CEA, CA19.9, Alpha Fetoprotein (AFP), PSA (Males)
11. Patients who are currently participating in another clinical study involving experimenting drugs and/or medical equipment.
12. Pregnant or Breastfeeding
13. Patients who are unable to perform the tests and assessments needed for the study
14. Patients who do not agree to participate in the study.
15. Patients with pre-morbid medical conditions, who have recently had alterations in their treatment regime (<6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2021-04-14 (Estimated); Study Completion 2022-04-14 (Estimated)

PRIMARY OUTCOMES:
To evaluate number of Participants with Treatment-Related Adverse Events | 1 year
  The safety of both Adipose derived and Umbilical Cord derived MSCs (both of Autologous and Allogenic sources) will be studied in clinical trial subjects. Adverse events will be documented and patients will be followed up over a period of 1 year post-infusion, to assess their well being. Clinical assessments and biochemical tests will be performed over the study period.
Improvement in General Well-Being, as assessed by our 'Quality of Life' Questionnaire, adapted from SF36. | 1 year
  A 'Quality of Life' Questionnaire will be filled by Trial Participants pre and post-infusion therapy. This questionnaire has been adapted from SF36 and scales of 1-5 are used to grade an individual's well being - A score of 1 being worse and 5 meaning a better outcome.
Change in inflammatory marker levels | 1 year
  IL-6, TNF alpha and CRP have been widely studied as markers of aging. These will be assessed in our trial subjects to ascertain if hMSC infusion results in any reduction in these inflammatory markers

SECONDARY OUTCOMES:
Change in medication dosage (if any) | 1 year
  IF patients with chronic medical conditions such as hypertension are on medication, patients will be assessed if hMSC infusion results in any change in required medication dosage

OTHER OUTCOMES:
Change from baseline, in plasma Glucose levels, over 52 weeks | 1 year
  fasting glucose levels and HbA1c Levels will be assessed pre and post-infusion
Fasting lipid profile | 1 year
  Fasting lipid profile will be assessed pre and post-infusion
Change in Hormonal Profile | 1 year
  FSH, LH, Estradiol, Progesterone, Testosterone Levels assessed pre and post-infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Landmark Medical Centre Sdn Bhd, Johor Bahru, Johor Darul Takzim, Malaysia